CLINICAL TRIAL: NCT01872364
Title: A Material Cost-Minimization Analysis for Hernia Repairs and Minor Procedures During a Surgical Mission in the Dominican Republic
Brief Title: Dominican Republic Mission Cost Analysis
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Jaime Cavallo, Postdoctorate Scholar, Washington University School of Medicine
Other Study IDs: 2013-05123
Record Dates: First submitted 2013-05-31; First posted 2013-06-07 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Hernia; Hydrocele
Keywords: Hernia repair; Hydrocelectomy; Global Health; Global Disease Burden; Surgical Mission; Dominican Republic; Cost-minimization; Procedural cost; Material cost; Item utilization; Excision of benign cutaneous mass; Minor procedure
MeSH Terms: conditions — Hernia; Testicular Hydrocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dominican Republic patients at NPO Outpatient Surgery Center

SUMMARY:
Expenditures on material supplies and medications constitute the greatest per capita costs for surgical missions. We hypothesized that supply acquisition at nonprofit organization cost would lead to significant cost-savings compared to supply acquisition at US academic institution costs from the provider perspective for hernia repairs and minor procedures during a surgical mission in the Dominican Republic.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Institute of Latin American Concern Center for surgical procedure, previously screened by local healthcare workers.
* Require hernia surgery, hydrocelectomy, excision of benign cutaneous mass.

Exclusion Criteria:

* Did not require hernia surgery, hydrocelectomy, excision of benign cutaneous mass.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to the Institute of Latin American Concern Center for surgical procedure, previously screened by local healthcare workers.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Expenditure on material supplies and medications | within 2 weeks
  Using quick response (QR) codes for accurate consumption accounting, non-profit and US academic institution unit costs are associated with each item in an electronic inventory system. Medication doses are recorded and QR codes for consumed items are scanned into a record for each sampled procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime A Cavallo, MD, MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Ozgediz D, Hsia R, Weiser T, Gosselin R, Spiegel D, Bickler S, Dunbar P, McQueen K. Population health metrics for surgery: effective coverage of surgical services in low-income and middle-income countries. World J Surg. 2009 Jan;33(1):1-5. doi: 10.1007/s00268-008-9799-y. PMID 18958518
- [Background] Taira BR, Kelly McQueen KA, Burkle FM Jr. Burden of surgical disease: does the literature reflect the scope of the international crisis? World J Surg. 2009 May;33(5):893-8. doi: 10.1007/s00268-009-9981-x. PMID 19290571
- [Background] Ozgediz D, Jamison D, Cherian M, McQueen K. The burden of surgical conditions and access to surgical care in low- and middle-income countries. Bull World Health Organ. 2008 Aug;86(8):646-7. doi: 10.2471/blt.07.050435. No abstract available. PMID 18797625
- [Background] Jamison DT, Breman JG, Measham AR, Alleyne G, Claeson M, Evans DB, Jha P, Mills A, Musgrove P, editors. Disease Control Priorities in Developing Countries. 2nd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK11728/ PMID 21250309
- [Background] Farmer PE, Kim JY. Surgery and global health: a view from beyond the OR. World J Surg. 2008 Apr;32(4):533-6. doi: 10.1007/s00268-008-9525-9. No abstract available. PMID 18311574
- [Background] Perkins RS, Casey KM, McQueen KA. Addressing the global burden of surgical disease: proceedings from the 2nd annual symposium at the American College of Surgeons. World J Surg. 2010 Mar;34(3):371-3. doi: 10.1007/s00268-009-0338-2. PMID 20041251
- [Background] McQueen KA, Hyder JA, Taira BR, Semer N, Burkle FM Jr, Casey KM. The provision of surgical care by international organizations in developing countries: a preliminary report. World J Surg. 2010 Mar;34(3):397-402. doi: 10.1007/s00268-009-0181-5. PMID 19685261
- [Background] Mock C, Cherian M, Juillard C, Donkor P, Bickler S, Jamison D, McQueen K. Developing priorities for addressing surgical conditions globally: furthering the link between surgery and public health policy. World J Surg. 2010 Mar;34(3):381-5. doi: 10.1007/s00268-009-0263-4. PMID 19876689
- [Background] Wang H, Dwyer-Lindgren L, Lofgren KT, Rajaratnam JK, Marcus JR, Levin-Rector A, Levitz CE, Lopez AD, Murray CJ. Age-specific and sex-specific mortality in 187 countries, 1970-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2071-94. doi: 10.1016/S0140-6736(12)61719-X. PMID 23245603
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Salomon JA, Vos T, Hogan DR, Gagnon M, Naghavi M, Mokdad A, Begum N, Shah R, Karyana M, Kosen S, Farje MR, Moncada G, Dutta A, Sazawal S, Dyer A, Seiler J, Aboyans V, Baker L, Baxter A, Benjamin EJ, Bhalla K, Bin Abdulhak A, Blyth F, Bourne R, Braithwaite T, Brooks P, Brugha TS, Bryan-Hancock C, Buchbinder R, Burney P, Calabria B, Chen H, Chugh SS, Cooley R, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, Davis A, Degenhardt L, Diaz-Torne C, Dorsey ER, Driscoll T, Edmond K, Elbaz A, Ezzati M, Feigin V, Ferri CP, Flaxman AD, Flood L, Fransen M, Fuse K, Gabbe BJ, Gillum RF, Haagsma J, Harrison JE, Havmoeller R, Hay RJ, Hel-Baqui A, Hoek HW, Hoffman H, Hogeland E, Hoy D, Jarvis D, Karthikeyan G, Knowlton LM, Lathlean T, Leasher JL, Lim SS, Lipshultz SE, Lopez AD, Lozano R, Lyons R, Malekzadeh R, Marcenes W, March L, Margolis DJ, McGill N, McGrath J, Mensah GA, Meyer AC, Michaud C, Moran A, Mori R, Murdoch ME, Naldi L, Newton CR, Norman R, Omer SB, Osborne R, Pearce N, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Pourmalek F, Prince M, Rehm JT, Remuzzi G, Richardson K, Room R, Saha S, Sampson U, Sanchez-Riera L, Segui-Gomez M, Shahraz S, Shibuya K, Singh D, Sliwa K, Smith E, Soerjomataram I, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Taylor HR, Tleyjeh IM, van der Werf MJ, Watson WL, Weatherall DJ, Weintraub R, Weisskopf MG, Whiteford H, Wilkinson JD, Woolf AD, Zheng ZJ, Murray CJ, Jonas JB. Common values in assessing health outcomes from disease and injury: disability weights measurement study for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2129-43. doi: 10.1016/S0140-6736(12)61680-8. PMID 23245605
- [Background] Salomon JA, Wang H, Freeman MK, Vos T, Flaxman AD, Lopez AD, Murray CJ. Healthy life expectancy for 187 countries, 1990-2010: a systematic analysis for the Global Burden Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2144-62. doi: 10.1016/S0140-6736(12)61690-0. PMID 23245606
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Pezzella AT. Volunteerism and humanitarian efforts in surgery. Curr Probl Surg. 2006 Dec;43(12):848-929. doi: 10.1067/j.cpsurg.2006.09.002. No abstract available. PMID 17222597
- [Background] Martiniuk AL, Manouchehrian M, Negin JA, Zwi AB. Brain Gains: a literature review of medical missions to low and middle-income countries. BMC Health Serv Res. 2012 May 29;12:134. doi: 10.1186/1472-6963-12-134. PMID 22643123
- [Background] Negus TL, Brown CJ, Konoske P. Determining medical staffing requirements for humanitarian assistance missions. Mil Med. 2010 Jan;175(1):1-6. doi: 10.7205/milmed-d-09-00051. PMID 20108835
- [Background] Hartgerink BJ, Chapman LE, Stevenson J, Donahue TF, Pagliara C. Utilization of surgical resources during the USNS COMFORT humanitarian mission to the Americas, June to October 2007. Mil Med. 2010 Sep;175(9):638-46. doi: 10.7205/milmed-d-09-00162. PMID 20882925
- [Background] Yeow VK, Lee ST, Lambrecht TJ, Barnett J, Gorney M, Hardjowasito W, Lemperle G, McComb H, Natsume N, Stranc M, Wilson L; International Task Force on Volunteer Cleft Missions. International Task Force on Volunteer Cleft Missions. J Craniofac Surg. 2002 Jan;13(1):18-25. doi: 10.1097/00001665-200201000-00003. PMID 11886986
- [Background] Gosselin RA, Maldonado A, Elder G. Comparative cost-effectiveness analysis of two MSF surgical trauma centers. World J Surg. 2010 Mar;34(3):415-9. doi: 10.1007/s00268-009-0230-0. PMID 19771466
- [Background] Moon W, Perry H, Baek RM. Is international volunteer surgery for cleft lip and cleft palate a cost-effective and justifiable intervention? A case study from East Asia. World J Surg. 2012 Dec;36(12):2819-30. doi: 10.1007/s00268-012-1761-3. PMID 22986629
- [Background] Turaga KK, Garg N, Coeling M, Smith K, Amirlak B, Jaszczak N, Elliott B, Manion J, Filipi C. Inguinal hernia repair in a developing country. Hernia. 2006 Aug;10(4):294-8. doi: 10.1007/s10029-006-0111-5. Epub 2006 Jul 19. PMID 16850136
- [Background] Shillcutt SD, Clarke MG, Kingsnorth AN. Cost-effectiveness of groin hernia surgery in the Western Region of Ghana. Arch Surg. 2010 Oct;145(10):954-61. doi: 10.1001/archsurg.2010.208. PMID 20956763
- [Background] Walk RM, Glaser J, Marmon LM, Donahue TF, Bastien J, Safford SD. Continuing promise 2009--assessment of a recent pediatric surgical humanitarian mission. J Pediatr Surg. 2012 Apr;47(4):652-7. doi: 10.1016/j.jpedsurg.2011.09.063. PMID 22498377
- [Background] Gil J, Rodriguez JM, Hernandez Q, Gil E, Balsalobre MD, Gonzalez M, Torregrosa N, Verdu T, Alcaraz M, Parrilla P. Do hernia operations in african international cooperation programmes provide good quality? World J Surg. 2012 Dec;36(12):2795-801. doi: 10.1007/s00268-012-1768-9. PMID 22976790
- [Background] Shillcutt SD, Sanders DL, Teresa Butron-Vila M, Kingsnorth AN. Cost-effectiveness of inguinal hernia surgery in northwestern Ecuador. World J Surg. 2013 Jan;37(1):32-41. doi: 10.1007/s00268-012-1808-5. PMID 23073503
- [Background] Mainthia R, Tye GW, Shapiro J, Doppenberg EM, Ward JD. A model for neurosurgical humanitarian aid based on 12 years of medical trips to South and Central America. J Neurosurg Pediatr. 2009 Jul;4(1):4-9. doi: 10.3171/2009.1.PEDS08193. PMID 19569901
- [Background] Doman DM, Blair JA, Napierala MA, Cho MS. Do plans and execution agree in a humanitarian medical mission? J Surg Orthop Adv. 2011 Spring;20(1):67-73. PMID 21477537
- [Background] Chen AT, Pedtke A, Kobs JK, Edwards GS Jr, Coughlin RR, Gosselin RA. Volunteer orthopedic surgical trips in Nicaragua: a cost-effectiveness evaluation. World J Surg. 2012 Dec;36(12):2802-8. doi: 10.1007/s00268-012-1702-1. PMID 22777413
- [Background] Ramirez-Fort MK, Lastra-Vicente R, Levitt JO, Sanchez JL, Reizner GT. Organizing a dermatology service mission. Int J Dermatol. 2013 Mar;52(3):342-9. doi: 10.1111/j.1365-4632.2012.05750.x. Epub 2012 Nov 1. PMID 23113920
- [Background] Maki J, Qualls M, White B, Kleefield S, Crone R. Health impact assessment and short-term medical missions: a methods study to evaluate quality of care. BMC Health Serv Res. 2008 Jun 2;8:121. doi: 10.1186/1472-6963-8-121. PMID 18518997
- [Background] Jha P, Bangoura O, Ranson K. The cost-effectiveness of forty health interventions in Guinea. Health Policy Plan. 1998 Sep;13(3):249-62. doi: 10.1093/heapol/13.3.249. PMID 10187595
- [Background] Uetani M, Jimba M, Niimi T, Natsume N, Katsuki T, Xuan le TT, Wakai S. Effects of a long-term volunteer surgical program in a developing country: the case in Vietnam from 1993 to 2003. Cleft Palate Craniofac J. 2006 Sep;43(5):616-9. doi: 10.1597/05-120. PMID 16986994
- [Background] Blanchard RJ, Merrell RC, Geelhoed GW, Ajayi OO, Laub DR, Rodas E. Training to serve unmet surgical needs worldwide. J Am Coll Surg. 2001 Oct;193(4):417-27. doi: 10.1016/s1072-7515(01)01037-7. No abstract available. PMID 11584970
- [Background] Welling DR, Ryan JM, Burris DG, Rich NM. Seven sins of humanitarian medicine. World J Surg. 2010 Mar;34(3):466-70. doi: 10.1007/s00268-009-0373-z. PMID 20063094
- [Background] Abenavoli FM. Improving humanitarian medical mission efficacy. Plast Reconstr Surg. 2012 Mar;129(3):559e-560e. doi: 10.1097/PRS.0b013e3182419a06. No abstract available. PMID 22374014
- [Background] Hilhorst D. Being good at doing good? Quality and accountability of humanitarian NGOs. Disasters. 2002 Sep;26(3):193-212. doi: 10.1111/1467-7717.00200. PMID 12227589
- [Background] Schneider WJ, Politis GD, Gosain AK, Migliori MR, Cullington JR, Peterson EL, Corlew DS, Wexler AM, Flick R, Van Beek AL. Volunteers in plastic surgery guidelines for providing surgical care for children in the less developed world. Plast Reconstr Surg. 2011 Jun;127(6):2477-2486. doi: 10.1097/PRS.0b013e3182131d2a. PMID 21311389
- [Background] Eberlin KR, Zaleski KL, Snyder HD, Hamdan US; Medical Missions for Children. Quality assurance guidelines for surgical outreach programs: a 20-year experience. Cleft Palate Craniofac J. 2008 May;45(3):246-55. doi: 10.1597/07-094.1. Epub 2008 Jan 1. PMID 18452366
- [Background] Hollier LH Jr, Sharabi SE, Koshy JC, Schafer ME, O'Young J, Flood TW. Surgical mission (not) impossible--now what? J Craniofac Surg. 2010 Sep;21(5):1488-92. doi: 10.1097/SCS.0b013e3181edc593. PMID 20818246
- See also: The World Factbook 2013 — https://www.cia.gov/library/publications/the-world-factbook/geos/dr.html
- See also: Smart traveler enrollment program (STEP). — https://step.state.gov/step/
- See also: Dominican Republic: country specific information — http://travel.state.gov/travel/cis_pa_tw/cis/cis_1103.html
- See also: Health information for travelers to the Dominican Republic — http://wwwnc.cdc.gov/travel/destinations/dominican-republic.htm